CLINICAL TRIAL: NCT05454345
Title: A Randomized Controlled Non-Inferiority Study for Shortening Tuberculosis Treatment With Sitafloxacin-Containing Regimens
Brief Title: Sitafloxacin-containing Regimens for Shortening Tuberculosis Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhang Ying, Prof, MD, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yzhang207
Record Dates: First submitted 2022-06-17; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — sitafloxacin; Trimethoprim, Sulfamethoxazole Drug Combination; Rifampin; Pyrazinamide; rifapentine; Isoniazid; Ethambutol; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin-containing regimen (Experimental): Thirteen weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and Sitafloxacin.
  Interventions: Drug: Sitafloxacin; Drug: Pyrazinamide; Drug: Rifapentine; Drug: Isoniazid
- The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin&SMZ/TMP-containing regimen (Experimental): Six weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and Sitafloxacin, followed by seven weeks of daily treatment with rifapentine, isoniazid, ,SMZ/TMP and Sitafloxacin.
  Interventions: Drug: Sitafloxacin; Drug: SMZ/TMP; Drug: Pyrazinamide; Drug: Rifapentine; Drug: Isoniazid
- The six-month standard Rifampin&Isoniazid&Pyrazinamide&Ethambutol-containing regimen (Active Comparator): Eight weeks of daily treatment with rifampin, isoniazid, pyrazinamide, and ethambutol, followed by Eighteen weeks of daily treatment with rifampin and isoniazid.
  Interventions: Drug: Rifampin; Drug: Pyrazinamide; Drug: Isoniazid; Drug: Ethambutol
- The four-month Rifapentine&Isoniazid&Pyrazinamide&Moxifloxacin -containing regimen (Active Comparator): Eight weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and moxifloxacin, followed by Nine weeks of daily treatment with rifapentine, isoniazid, and moxifloxacin.
  Interventions: Drug: Rifapentine; Drug: Isoniazid; Drug: Ethambutol; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Sitafloxacin — In our Intervention group, sitafloxacin replace the ethambutol, 200mg/d
  Arms: The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin&SMZ/TMP-containing regimen; The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin-containing regimen
Drug: SMZ/TMP — In our The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin&SMZ/TMP-containing regimen, Six weeks of daily treatment with rifapentine, isoniazid, pyrazinamide, and Sitafloxacin, followed by seven weeks of daily treatment with rifapentine, isoniazid, ,SMZ/TMP and Sitafloxacin, SMZ 80mg/kg/d, TMP16mg/kg/d
  Arms: The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin&SMZ/TMP-containing regimen
Drug: Rifampin — Rifampin is a first-line antimicrobial agent against drug-susceptible tuberculosis in WHO guideline, Rifampin 600mg (8-12mg/kg/d)
  Arms: The six-month standard Rifampin&Isoniazid&Pyrazinamide&Ethambutol-containing regimen
Drug: Pyrazinamide — Pyrazinamide is a first-line antimicrobial agent against drug-susceptible tuberculosis in WHO guideline, 2000mg (20-30mg/kg/d)
  Arms: The six-month standard Rifampin&Isoniazid&Pyrazinamide&Ethambutol-containing regimen; The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin&SMZ/TMP-containing regimen; The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin-containing regimen
Drug: Rifapentine — In our Intervention group, rifapentine replace rifampin, 600mg/d
  Arms: The four-month Rifapentine&Isoniazid&Pyrazinamide&Moxifloxacin -containing regimen; The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin&SMZ/TMP-containing regimen; The three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin-containing regimen
Drug: Isoniazid — Isoniazid is a first-line antimicrobial agent against drug-susceptible tuberculosis in WHO guideline, 300mg (4-6mg/kg/d)
Drug: Ethambutol — Ethambutol is a first-line antimicrobial agent against drug-susceptible tuberculosis in WHO guideline, 1200mg (15-25mg/kg/d)
  Arms: The four-month Rifapentine&Isoniazid&Pyrazinamide&Moxifloxacin -containing regimen; The six-month standard Rifampin&Isoniazid&Pyrazinamide&Ethambutol-containing regimen
Drug: Moxifloxacin — Moxifloxacin is a fourth-generation fluoroquinolone with potent activity against M. tuberculosis in vitro and in vivo, 400mg (7.5-10mg/kg/d)
  Arms: The four-month Rifapentine&Isoniazid&Pyrazinamide&Moxifloxacin -containing regimen

SUMMARY:
This study is a clinical trial conducted to determine whether the sitafloxacin-containing three-month regimens are as effective as the standard six-month regimen and the four-month rifapentine and moxifloxacin regimen (substitution of rifapentine for rifampin and moxifloxacin for ethambutol) for treatment of pulmonary tuberculosis. The standard six-month regimen is two months of isoniazid, rifampin, ethambutol, and pyrazinamide, followed by four months of isoniazid and rifampin. The four-month regimen consists of two months of isoniazid, rifapentine, moxifloxacin, and pyrazinamide, followed by two months of isoniazid rifapentine and moxifloxacin. The new three-month tuberculosis treatment regimens are six weeks of isoniazid, rifapentine, Sitafloxacin, and pyrazinamide, followed by seven weeks of isoniazid, rifapentine, and Sitafloxacin, or 13 weeks of isoniazid, rifapentine, Sitafloxacin, and pyrazinamide. The primary research question is to evaluate the efficacy and safety of the 3 month Sitafloxacin-containing regimen, and to determine if it can shorten the treatment of drug-susceptible pulmonary tuberculosis while achieving non-inferiority in treatment success with the current 6 month and 4 month treatment regimens. Safety, side effects of Sitafloxacin for participants in the clinical trial are also assessed. Rates of cure, treatment success, recurrence, and cure (cure without recurrence) are determined for subgroup analysis in the standard six-month regimen group, the four-month regimen group, and two three-month regimen groups.

DETAILED DESCRIPTION:
1. TB disease-free survival at 13 weeks after study treatment assignment among participants in the three-month regimen group 1 and 2, the four-month regimen group, and the standard six-month regimen. The patients are AFB sputum smear negative or culture negative for M. tuberculosis, two assays are performed (each test is separated by at least seven days), eliminating the M. tuberculosis load from a pulmonary infection.
2. Persons with positive culture results for M. tuberculosis or smear-positive sputum(spoligotyping isolates genetically identified as M. tuberculosis).
3. Data collected pre-study included written informed consent; patients assessed for eligibility; height and weight; clinical symptoms of TB; adjunctive therapy; adverse drug reaction; blood and urine routine; liver and kidney function; acid-fast staining; single M. tuberculosis strain isolated from one patient with TB; GeneXpert MTB/RIF; chest CT scans
4. Clinical symptoms of TB: cough, expectoration, hemoptysis, chest pain, fever, shortness of breath, weak.
5. All patients should review for Xpert MTB/RIF assay in the second week.
6. During treatment, clinical symptoms of TB and body weights takes weekly; blood and urine routine in weeks 1,2,4,8,13; Sputum smears and culture were routinely in weeks 1,2,4,8,13, and months 6 and 12. TB Disease-free Survival at six or twelve months after study treatment assignment as the secondary outcome measures.
7. TB patients were identified through bacteriological confirmation (smear-positive and/or culture-positive).
8. Pulmonary TB patients showed manifestation of tuberculosis by chest CT scans or X-ray.
9. Adverse events of the treatment: neurological diseases, blood system diseases; diseases of the circulatory system; respiratory diseases; digestive diseases; extra-pulmonary TB; diabetes; arthralgia; mental disorders; hemoptysis and pneumothorax; pulmonary embolism; skin rash.
10. Management of a participant with a positive sputum culture for M. tuberculosis at or after week 13: A second sputum sample was collected on the following day for a second culture. If M. tuberculosis is isolated in culture, drug susceptibility testing should be performed on one isolate. Patients will re-evaluate symptoms and chest CT scans; sputum was performed in triplicates and repeated for validation. These patients could restart the standard six-month regimen at any time.
11. Patients follow up one week after the completion of treatment and 6,12,18 months after treatment is over. Patients undergo regular follow-up with sputum smear tests or imaging studies. Patients with positive TB symptom screen or suspected TB patients based on imaging tests are recommended with research staff.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years to 70.
2. At least one sputum specimen is positive for acid-fast bacilli or positive results of sputum culture on smear microscopy(species identification as M. tuberculosis) or at least one sputum specimen positive for M. tuberculosis by Xpert MTB/RIF testing.
3. Phenotypic drug susceptibility testing indicates the patient's isolate is susceptible to rifampin, isoniazid, pyrazinamide, ethambutol, rifapentine, moxifloxacin, and Sitafloxacin.
4. Patients have written informed consent.

Exclusion Criteria:

1. Extra-pulmonary or Disseminated TB.
2. HIV-positive individuals, steroid-dependent and those on steroid treatment.
3. Autoimmune diseases, severe hepatic or renal dysfunction, psychosis, hematological malignancies, cancer, diabetes individuals.
4. Known allergy to one or more of the study drugs.
5. Women who are currently pregnant or breast-feeding.
6. Patients who received any investigational drug in the past three months.
7. The patients refused treatment with medications
8. Mycobacterium tuberculosis/nontuberculous mycobacterium co-infection.
9. In the investigator's judgment, other medical conditions that are not in the individual's best interest to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
TB Disease-free Survival after the completion of the treatment cycle. | Week 13 in the three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin-containing regimen and three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin&SMZ/TMP-containing regimen
  To evaluate the efficacy of a Sitafloxacin-containing regimen to determine whether the substitution of Sitafloxacin for moxifloxacin could shorten the treatment duration from 6 months to 3 months (13 weeks) for drug-susceptible pulmonary tuberculosis. Pathogen detection (including sputum smear and sputum culture) should complete in Week 13 in the three-month regimen group, Week 17 in the four-month regimen group, and Week 26 in the standard six-month regimen group.
TB Disease-free Survival after the completion of the treatment cycle. | Week 17 in the four-month Rifapentine&Isoniazid&Pyrazinamide&Moxifloxacin -containing regimen
  To evaluate the efficacy of a Sitafloxacin-containing regimen to determine whether the substitution of Sitafloxacin for moxifloxacin could shorten the treatment duration from 6 months to 3 months (13 weeks) for drug-susceptible pulmonary tuberculosis. Pathogen detection (including sputum smear and sputum culture) should complete in Week 13 in the three-month regimen group, Week 17 in the four-month regimen group, and Week 26 in the standard six-month regimen group.
TB Disease-free Survival after the completion of the treatment cycle. | Week 26 in the six-month standard Rifampin&Isoniazid&Pyrazinamide&Ethambutol-containing regimen
  To evaluate the efficacy of a Sitafloxacin-containing regimen to determine whether the substitution of Sitafloxacin for moxifloxacin could shorten the treatment duration from 6 months to 3 months (13 weeks) for drug-susceptible pulmonary tuberculosis. Pathogen detection (including sputum smear and sputum culture) should complete in Week 13 in the three-month regimen group, Week 17 in the four-month regimen group, and Week 26 in the standard six-month regimen group.
Percentage Participants With Grade 3 or Higher Adverse Events During Study Drug Treatment in Control Regimen | Week 13 in the three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin-containing regimen and three-month Rifapentine&Isoniazid&Pyrazinamide&Sitafloxacin&SMZ/TMP-containing regimen
  To determine Grade 3 or higher adverse events in study participants during drug treatment in the standard six-month regimen, the four-month regimen, and the three-month regimen Sitafloxacin-containing and three-month Sitafloxacin&SMZ/TMP-containing regimen
Percentage Participants With Grade 3 or Higher Adverse Events During Study Drug Treatment in Control Regimen | Week 17 in the four-month Rifapentine&Isoniazid&Pyrazinamide&Moxifloxacin -containing regimen
  To determine Grade 3 or higher adverse events in study participants during drug treatment in the standard six-month regimen, the four-month regimen, and the three-month regimen Sitafloxacin-containing and three-month Sitafloxacin&SMZ/TMP-containing regimen
Percentage Participants With Grade 3 or Higher Adverse Events During Study Drug Treatment in Control Regimen | Week 26 in the six-month standard Rifampin&Isoniazid&Pyrazinamide&Ethambutol-containing regimen
  To determine Grade 3 or higher adverse events in study participants during drug treatment in the standard six-month regimen, the four-month regimen, and the three-month regimen Sitafloxacin-containing and three-month Sitafloxacin&SMZ/TMP-containing regimen

SECONDARY OUTCOMES:
The rates of negative sputum conversion | two months
  The rates of negative sputum conversion will be determined at the end of 2 months using the sputum smear and culture test.
TB disease-free survival at six and twelve months after study treatment assignment. | Twelve months
  The rates of TB disease-free survival at six and twelve months

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Guidelines for the Programmatic Management of Drug-Resistant Tuberculosis: 2011 Update. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK148644/ PMID 23844450
- [Background] Gupta VK, Kumar MM, Singh D, Bisht D, Sharma S. Drug targets in dormant Mycobacterium tuberculosis: can the conquest against tuberculosis become a reality? Infect Dis (Lond). 2018 Feb;50(2):81-94. doi: 10.1080/23744235.2017.1377346. Epub 2017 Sep 21. PMID 28933243
- [Background] Burman WJ, Gallicano K, Peloquin C. Comparative pharmacokinetics and pharmacodynamics of the rifamycin antibacterials. Clin Pharmacokinet. 2001;40(5):327-41. doi: 10.2165/00003088-200140050-00002. PMID 11432536
- [Background] Dorman SE, Nahid P, Kurbatova EV, Phillips PPJ, Bryant K, Dooley KE, Engle M, Goldberg SV, Phan HTT, Hakim J, Johnson JL, Lourens M, Martinson NA, Muzanyi G, Narunsky K, Nerette S, Nguyen NV, Pham TH, Pierre S, Purfield AE, Samaneka W, Savic RM, Sanne I, Scott NA, Shenje J, Sizemore E, Vernon A, Waja Z, Weiner M, Swindells S, Chaisson RE; AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Four-Month Rifapentine Regimens with or without Moxifloxacin for Tuberculosis. N Engl J Med. 2021 May 6;384(18):1705-1718. doi: 10.1056/NEJMoa2033400. PMID 33951360
- [Background] Keating GM. Sitafloxacin: in bacterial infections. Drugs. 2011 Apr 16;71(6):731-44. doi: 10.2165/11207380-000000000-00000. PMID 21504249
- [Background] Yamaguchi K, Ohno A, Ishii Y, Tateda K, Iwata M, Kanda M, Akizawa K, Shimizu C, Kon S, Nakamura K, Matsuda K, Tominaga M, Nakagawa T, Sugita A, Ito T, Kato J, Suwabe A, Yamahata K, Kawamura C, Tashiro H, Horiuchi H, Katayama Y, Kondou S, Misawa S, Murata M, Kobayashi Y, Okamoto H, Yamazaki K, Okada M, Haruki K, Kanno H, Aihara M, Maesaki S, Hashikita G, Miyajima E, Sumitomo M, Saito T, Yamane N, Kawashima C, Akiyama T, Ieiri T, Yamamoto Y, Okamoto Y, Okabe H, Moro K, Shigeta M, Yoshida H, Yamashita M, Hida Y, Takubo T, Kusakabe T, Masaki H, Heijyou H, Nakaya H, Kawahara K, Sano R, Matsuo S, Kono H, Yuzuki Y, Ikeda N, Idomuki M, Soma M, Yamamoto G, Kinoshita S, Kawano S, Oka M, Kusano N, Kang D, Ono J, Yasujima M, Miki M, Hayashi M, Okubo S, Toyoshima S, Kaku M, Sekine I, Shiotani J, Horiuchi H, Tazawa Y, Yoneyama A, Kumasaka K, Koike K, Taniguchi N, Ozaki Y, Uchida T, Murakami M, Inuzuka K, Gonda H, Yamaguchi I, fujimoto Y, Iriyama J, Asano Y, Genma H, Maekawa M, Yoshimura H, Nakatani K, Baba H, Ichiyama S, Fujita S, Kuwabara M, Okazaki T, Fujiwara H, Ota H, Nagai A, Fujita J, Negayama K, Sugiura T, Kamioka M, Murase M, Yamane N, Nakasone I, Okayama A, Aoki Y, Kusaba K, Nakashima Y, Miyanohara H, Hiramatsu K, Saikawa T, Yanagihara K, Matsuda J, Kohno S, Mashiba K. [In vitro susceptibilities to levofloxacin and various antibacterial agents of 12,919 clinical isolates obtained from 72 centers in 2007]. Jpn J Antibiot. 2009 Aug;62(4):346-70. Japanese. PMID 19860322
- [Background] Asakura T, Suzuki S, Fukano H, Okamori S, Kusumoto T, Uwamino Y, Ogawa T, So M, Uno S, Namkoong H, Yoshida M, Kamata H, Ishii M, Nishimura T, Hoshino Y, Hasegawa N. Sitafloxacin-Containing Regimen for the Treatment of Refractory Mycobacterium avium Complex Lung Disease. Open Forum Infect Dis. 2019 Mar 7;6(4):ofz108. doi: 10.1093/ofid/ofz108. eCollection 2019 Apr. PMID 31111076
- [Background] Ito S, Yasuda M, Seike K, Sugawara T, Tsuchiya T, Yokoi S, Nakano M, Deguchi T. Clinical and microbiological outcomes in treatment of men with non-gonococcal urethritis with a 100-mg twice-daily dose regimen of sitafloxacin. J Infect Chemother. 2012 Jun;18(3):414-8. doi: 10.1007/s10156-012-0392-9. Epub 2012 Feb 28. PMID 22370921
- [Background] Mori H, Suzuki H, Matsuzaki J, Masaoka T, Kanai T. 10-Year Trends in Helicobacter pylori Eradication Rates by Sitafloxacin-Based Third-Line Rescue Therapy. Digestion. 2020;101(5):644-650. doi: 10.1159/000501610. Epub 2019 Aug 6. PMID 31387107
- [Background] Li Y, Zhu D, Peng Y, Tong Z, Ma Z, Xu J, Sun S, Tang H, Xiu Q, Liang Y, Wang X, Lv X, Dai Y, Zhu Y, Qu Y, Xu K, Huang Y, Wu S, Lai G, Li X, Han X, Yang Z, Sheng J, Liu Z, Li H, Chen Y, Zhu H, Zhang Y. A randomized, controlled, multicenter clinical trial to evaluate the efficacy and safety of oral sitafloxacin versus moxifloxacin in adult patients with community-acquired pneumonia. Curr Med Res Opin. 2021 Apr;37(4):693-701. doi: 10.1080/03007995.2021.1885362. Epub 2021 Feb 22. PMID 33534617
- [Background] Leechawengwongs M, Prammananan T, Jaitrong S, Billamas P, Makhao N, Thamnongdee N, Thanormchat A, Phurattanakornkul A, Rattanarangsee S, Ratanajaraya C, Disratthakit A, Chaiprasert A. In Vitro Activity and MIC of Sitafloxacin against Multidrug-Resistant and Extensively Drug-Resistant Mycobacterium tuberculosis Isolated in Thailand. Antimicrob Agents Chemother. 2017 Dec 21;62(1):e00825-17. doi: 10.1128/AAC.00825-17. Print 2018 Jan. PMID 29061759
- [Background] Kamada K, Yoshida A, Iguchi S, Arai Y, Uzawa Y, Konno S, Shimojima M, Kikuchi K. Nationwide surveillance of antimicrobial susceptibility of 509 rapidly growing mycobacteria strains isolated from clinical specimens in Japan. Sci Rep. 2021 Jun 9;11(1):12208. doi: 10.1038/s41598-021-91757-4. PMID 34108590
- [Background] Yi L, Aono A, Chikamatsu K, Igarashi Y, Yamada H, Takaki A, Mitarai S. In vitro activity of sitafloxacin against Mycobacterium tuberculosis with gyrA/B mutations isolated in Japan. J Med Microbiol. 2017 Jun;66(6):770-776. doi: 10.1099/jmm.0.000493. PMID 28598311
- [Background] Suzuki Y, Nakajima C, Tamaru A, Kim H, Matsuba T, Saito H. Sensitivities of ciprofloxacin-resistant Mycobacterium tuberculosis clinical isolates to fluoroquinolones: role of mutant DNA gyrase subunits in drug resistance. Int J Antimicrob Agents. 2012 May;39(5):435-9. doi: 10.1016/j.ijantimicag.2012.01.007. Epub 2012 Mar 13. PMID 22421328
- See also: WHO guideline — https://www.who.int/publications-detail-redirect/9789241550529